CLINICAL TRIAL: NCT00637949
Title: A 6-Week Multicenter, Randomized, Double-Blind, Double-Dummy, Active-Controlled Parallel Group Clinical Saftey Study to Evaluate Incidence of Predefined Gastrointestinal Adverse Events and Peripheral Edema in Subjects With Primary Osteoarthritis Treated With COX189 400 mg o-do Using Rofecoxib 25 mg o.d. as a Comparator
Brief Title: Safety of Lumiracoxib in Patients With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2307
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; lumiracoxib; rofecoxib; Cox-2; Osteoarthritis (primary osteoarthritis hip, hand, knee or spine (cervical or lumbar)
MeSH Terms: conditions — Osteoarthritis | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Device: lumiracoxib
- 2 (Active Comparator)
  Interventions: Drug: rofecoxib

INTERVENTIONS:
Device: lumiracoxib — 400 mg once daily, oral over 6 weeks
  Other Names: Prexige
  Arms: 1
Drug: rofecoxib — 25 mg, oral, daily over 6 weeks
  Other Names: Vioxx
  Arms: 2

SUMMARY:
This safety study evaluated the incidence of gastrointestinal adverse events and edema in patients with osteoarthritis treated with lumiracoxib and rofecoxib as comparator

ELIGIBILITY:
Inclusion Criteria:

* Age >=50 years old
* Primary osteoarthritis in hip, hand, knee or spine for at least 3 month
* Pain in the target joint of moderate intensity
* Written informed consent

Exclusion Criteria:

* Secondary osteoarthritis
* Active upper gastro intestinal tract ulceration
* Inflammatory joint disease
* Gout
* Clinically significant hepatic or renal disease

Other in and exclusion criteria may apply

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2000-12; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Incidence of at least one of seven predefined gastrointestinal adverse events | 6 weeks

REFERENCES:
- [Derived] Stricker K, Yu S, Krammer G. A 6-week, multicentre, randomised, double-blind, double-dummy, active-controlled, clinical safety study of lumiracoxib and rofecoxib in osteoarthritis patients. BMC Musculoskelet Disord. 2008 Sep 8;9:118. doi: 10.1186/1471-2474-9-118. PMID 18778469